CLINICAL TRIAL: NCT05478564
Title: INTRAOPERATIVE HEMODYNAMIC MANAGEMENT IN ABDOMINAL AORTIC SURGERY GUIDED BY HYPOTENSION PREDICTION INDEX (HPI) - HEMAS Trial
Brief Title: Hemodynamic Monitoring During Abdominal Aortic Surgery
Acronym: HEMAS
Status: Completed | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Enrico Giustiniano, Dr, Humanitas Clinical and Research Center
Other Study IDs: HEMAS; 3236 (Other: Ethical Committee authorization)
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2022-11

CONDITIONS: Hemodynamic Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Intraoperative fluids and vasoactive drugs management protocol — Limitation of hypotensive events during open surgery for abdominal aorta repair
  Other Names: In case of >20% ignored protocol (poor adherence), patient will be excluded

SUMMARY:
This trial investigates the ability of our istitutional algorithm in maintaining a safe hemodynamics during abdominal aorta open surgery, in terms of limitation of intraoperative hypotension incidence

DETAILED DESCRIPTION:
The present trial includes patients submitted to abdominal aorta open surgery. This type of procedure is very challenging for the hemodynamic management because of the operation per se (during which the surgeon clamp and unclamp the aorta with very significant hemodynamic variations) and because of the altered tone of the vessels due to the general vascular disease such a type of patients is suffering from.

The aim of this study is to verify if the incidence of intraoperative hypotension in terms of severity, lasting and number of episodes, may be reduced by the application of a protocol of hemodynamic management.

Primary endpoint: Global time spent in hypotension <10%.

Secondary Endpoints:

1. Time Weighted Average (TWA) of Area Under the Threshold <0.4 mmHg
2. Incidence of hypotensive events/patient < 8 (including the expected hypotensive events due to the aortic clamping and unclamping)

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoing abdominal aorta open surgical repair

Exclusion Criteria:

* Emergent/urgent operation
* Age <18 years
* Pregnancy
* Intra-operative blood loss > or = 3000ml

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults submitted to open surgery due to abdominal aorta repair
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Global time spent in hypotension <10% | Intraoperative period
  Hypotension=mean arterial pressure <65 mmHg for at least 1 minute

SECONDARY OUTCOMES:
Time Weighted Average (TWA) of Area Under the Threshold <0.4 mmHg | Intraoperative period
  The severity of hypotension during the whole intraoperative surgery
Incidence of hypotensive events/patient < 8 | Intraoperative period
  including the expected hypotensive events due to the aortic clamping and unclamping

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Clinical and Research center, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giustiniano E, Nisi F, Ferrod F, Lionetti G, Viscido C, Reda A, Piccioni F, Buono G, Cecconi M. Intraoperative hemodynamic management in abdominal aortic surgery guided by the Hypotension Prediction Index: the Hemas multicentric observational study. J Anesth Analg Crit Care. 2025 Feb 13;5(1):7. doi: 10.1186/s44158-024-00222-x. PMID 39948674